CLINICAL TRIAL: NCT04009668
Title: Precision Medicine Proof of Concept for Tumor Necrosis Factor Inhibition in Focal Segmental Glomerulosclerosis and Treatment Resistant Minimal Change Disease
Brief Title: Tumor Necrosis Factor Inhibition in Focal Segmental Glomerulosclerosis and Treatment Resistant Minimal Change Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Zubin Juzer Modi, Assistant Professor of Pediatrics, Division of Nephrology, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HUM00147018
Record Dates: First submitted 2019-07-02; First posted 2019-07-05 (Actual); Results first posted 2024-10-30 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: FSGS; MCD; Focal Segmental Glomerulosclerosis; Minimal Change Disease
Keywords: Kidney Disease; Minimal Change Disease; Nephrotic Syndrome; Focal Segmental Glomerulosclerosis; FSGS
MeSH Terms: conditions — Macular dystrophy, corneal type 1; Glomerulosclerosis, Focal Segmental; Nephrosis, Lipoid; Kidney Diseases; Nephrotic Syndrome | interventions — Adalimumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- adalimumab (Experimental): Adalimumab dose every other week (study weeks 0, 2, 4, 6, and 8), subcutaneously
  Interventions: Drug: adalimumab

INTERVENTIONS:
Drug: adalimumab — Adalimumab will be dosed based on weight
  Other Names: Humira

SUMMARY:
Adalimumab, a treatment which blocks tumor necrosis factor (TNF), was tested to see if it changed levels of urine biomarker levels, tissue inhibitor of metalloprotease-1 (TIMP1), and monocyte chemoattractant protein-1 (MCP1). Results may help develop individualized treatment options for future patients with TNF-driven focal segmental glomerulosclerosis (FSGS) or minimal change disease (MCD).

ELIGIBILITY:
Inclusion Criteria:

* Kidney biopsy confirmed Focal Segmental Glomerulosclerosis (FSGS) or Minimal Change Disease (MCD)
* For Minimal Change Disease patients only, history of resistance to corticosteroid therapy
* Increased urinary excretion of biomarkers of Tumor Necrosis Factor (TNF) activation (MCP1/Cr and/ or TIMP1/Cr) at study screening
* eGFR>30 ml/min/1.73 m2 at screening
* Urine protein:creatinine ratio ≥1.5 g/g at screening
* Weight >15 kg
* Stable therapy with angiotensin converting enzyme inhibitors, angiotensin receptor blockers, and oral immunosuppression agents for at least 30 days prior to enrollment
* Birth control use in females of child bearing potential
* Informed consent and assent if applicable

Exclusion Criteria:

* Kidney or other solid organ or bone marrow transplant recipient
* Allergy or intolerance to investigational agent
* Secondary Focal Segmental Glomerulosclerosis (FSGS)
* Severe obesity
* Live virus vaccine in the past 3 months
* Malignancy, current or in the past 5 years
* Active local or systemic bacterial, fungal or viral infection
* Active or latent Hepatitis B, Hepatitis C, HIV, or tuberculosis
* History of demyelinating disease, e.g. Multiple Sclerosis or Guillain-Barre
* History of heart failure
* Active liver disease
* Systemic lupus erythematosus or ANA > 1:80
* History of inflammatory bowel disease, e.g. ulcerative colitis or Crohns disease
* Cyclophosphamide in past 90 days, Rituximab in the past 180 days
* Pregnancy or nursing
* Blood white blood cell count <4,500/mm3; Hg <9 g/dL; Platelet count <150,000/mm3 at enrollment. - Use of an erythropoiesis stimulating agent will not be an exclusion criterion.
* Concurrent use of interleukin-1 antagonist (Anakinra), other TNF blocking agent, methotrexate or abatacept
* Diabetes Mellitus

Ages: 6 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-10-02 (Actual); Primary Completion 2023-09-05 (Actual); Study Completion 2023-10-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zubin Modi, MD, Study Director — University of Michigan
Locations (4):
- United States (4):
  - The University of Michigan, Ann Arbor, Michigan
  - New York University, New York, New York
  - Levine Children's Hospital/Atrium Health, Charlotte, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: Yes
This trial will follow the publication and data sharing policies of the NEPTUNE study, www.NEPTUNE-study.org
  Request for ancillary studies should be submitted through the project contact and will be reviewed by the project steering committee.
  After the study is completed, data will be submitted to the Nephrotic Syndrome Study Network (NEPTUNE), an NIH funded consortium. Proposals to access the data will then be submitted via the NEPTUNE Ancillary Studies program (NEPTUNE-study.org). Following closure of NEPTUNE, the trial data will convey with the NEPTUNE date to the NIH/NIDDK repository and can be accessed through this mechanism following approval.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: At the latest, data will be shared with the NEPTUNE Data Analysis and Coordinating Center at the time of publication of final results or 24 months after transfer of samples or raw data sets.
Access Criteria: While this study is open data requests from this study will need to seek approval from the trial steering committee.
  Once the data is transferred to the NEPTUNE study, all study data will become part of the aggregate NEPTUNE data and available to NEPTUNE participant sites and other requesting third parties upon request. Subsequent access to these data will be governed by the NIH Office of Rare Diseases (ORD) data sharing policies.
URL: http://neptune-study.org/

REFERENCES:
- [Derived] Trachtman H, Modi ZJ, Ju W, Lee E, Chinnakotla S, Massengill S, Sedor J, Mariani L, Zhai Y, Hao W, Desmond H, Eddy S, Ramani K, Spino C, Kretzler M. Precision Medicine Proof-of-Concept Study of a TNF Inhibitor in FSGS and Treatment-Resistant Minimal Change Disease. Kidney360. 2025 Feb 1;6(2):284-295. doi: 10.34067/KID.0000000635. Epub 2024 Nov 18. PMID 39808779

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: 2019-2023 Recruitment Sites: University of Michigan, Ann Arbor, MI; New York University Langone Health, New York, NY; Cleveland Clinic, Cleveland, OH; Levine Children's Hospital at Atrium Health, Charlotte, NC.
Pre-assignment Details: Following consent, participants provided a urine sample to measure urinary monocyte chemoattractant protein-1 (uMCP-1) and urinary tissue inhibitor of metalloprotease-1 (uTIMP-1), two indicators of intra-renal tumor necrosis factor (TNF) pathway activation. Participants with present TNF activation were advanced to screening. Upon confirmation of eligibility, participants proceeded to the treatment phase.
Groups:
- Adalimumab: Adalimumab dose every other week (study weeks 0, 2, 4, 6, and 8), subcutaneously. Adalimumab will be dosed based on weight (20 mg for subjects weighing 15kg to <30kg, or 40 mg for subjects >30kg).
Period: Overall Study
Arm/Group | Adalimumab
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Adalimumab
Number analyzed (Participants) | 7
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 15.9 [12.8 to 19.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black or African American | 1
  Race: Native Hawaiian or Other Pacific Islander | 1
  Race: White | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 3
  Ethnicity: Not Hispanic or Latino | 4
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Change in Urine MCP1/Cr Levels
Description: MCP1 is an established marker of intra-renal TNF pathway activation. A reduction in MCP1 reflects a reduction in the activation of the TNF pathway in the kidney. Values were measured by enzyme-linked immunosorbent assay (ELISA) testing and standardized over serum creatinine.
Time Frame: 10 Weeks
Measure: Median (Inter-Quartile Range); unit: ng/mg
Arm/Group | Adalimumab
Number analyzed (Participants) | 7
ng/mg
  Baseline | 5.57 [0.79 to 6.61]
  Week 10 | 2.89 [1.36 to 7.14]

2. Primary Outcome: Change in Urine TIMP1/Cr Levels
Description: TIMP1 is an established marker of intra-renal TNF pathway activation. A reduction in TIMP1 reflects a reduction in the activation of the TNF pathway in the kidney. Values were measured by enzyme-linked immunosorbent assay (ELISA) testing and standardized over serum creatinine.
Time Frame: 10 Weeks
Measure: Median (Inter-Quartile Range); unit: ng/mg
Arm/Group | Adalimumab
Number analyzed (Participants) | 7
ng/mg
  Baseline | 41.34 [3.64 to 75.38]
  Week 10 | 31.36 [4.39 to 146.86]

3. Secondary Outcome: Incidence of Adverse Events (AEs)
Description: AEs for this outcome measure were classified using the following definitions:
  * Mild: no or mild symptoms, and not requiring intervention
  * Moderate: with minimal or local intervention, and limiting age-appropriate activities
  * Severe: intervention necessary and limiting age-appropriate activities but not immediately life-threatening, and requiring hospitalization or prolongation of hospitalization
  * Serious AE: results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability/incapacity, pregnancy or congenital anomaly/birth defect.
  Some participants experienced multiple types of AE during the course of the trial.
Time Frame: 14 weeks
Measure: Number; unit: Adverse Event
Arm/Group | Adalimumab
Number analyzed (Participants) | 7
Adverse Event
  Mild AEs | 7
  Moderate AEs | 4
  Severe AEs | 1
  Serious AEs | 10

4. Secondary Outcome: Change in Estimated Glomerular Filtration Rate (eGFR)
Description: eGFR is a measure of kidney functioning based on a blood sample and clinical information to calculate it. Normal kidney function is greater than 90 ml/min/1.73 m2. Result data is the percent change in eGFR following the intervention. The lower the number shows the greater decline in kidney function.
Time Frame: 10 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | Adalimumab
Number analyzed (Participants) | 7
Percent Change | -28.90 [-30.50 to -12.18]

5. Secondary Outcome: Change in Urine Protein Creatinine Ratio (UPCR)
Description: UPCR is a measure of protein spillage from the kidney based on a urine specimen. Normal reference range is less than 0.03 mg/mg. Result is the percent change in UPCR following the intervention, with lower number showing less protein spilling from the kidney, reflecting better disease control.
Time Frame: 10 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | Adalimumab
Number analyzed (Participants) | 7
Percent Change | -11.60 [-23.45 to -9.28]

6. Secondary Outcome: Proportion of Participants Who Achieved Both a Nadir Urine Protein Creatinine Ratio (UPCR) of Less Than 1.5 g/g and at Least a 40% Reduction From Baseline
Description: UPCR is a measure of protein spillage from the kidney based on a urine specimen. Normal reference range is less than 0.03 mg/mg. Result is the count of participants who simultaneously met the criteria of having both a raw UPCR value of less than 1.5 g/g and at least a 40% reduction from baseline.
Time Frame: 10 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 7
Participants | 2

ADVERSE EVENTS:
Time Frame: 14 Weeks
Arm/Group | Adalimumab
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 1/7
Other Adverse Events (participants affected / at risk) | 5/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adalimumab (N=7)
Influenza (Infections and infestations) | 1 (1)
Edema (Renal and urinary disorders) | 1 (5)
Anasarca and AKI (Renal and urinary disorders) | 1 (4)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adalimumab (N=7)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Volume depletion (General disorders) | 1 (1)
COVID-19 (Infections and infestations) | 2 (2)
Rhinovirus (Infections and infestations) | 1 (1)
Increased edema (Renal and urinary disorders) | 1 (1)
eGFR decline (greater than 25% since baseline) (Renal and urinary disorders) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Recruitment was launched in Dec. 2019 and was significantly impacted by the COVID-19 pandemic with most participants enrolling in 2022.

One participant was unable to attend the week 10 visit because of COVID-19 infection, and the week 8 biomarker results were used to determine the primary outcome.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2023-02-21): https://cdn.clinicaltrials.gov/large-docs/68/NCT04009668/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-31): https://cdn.clinicaltrials.gov/large-docs/68/NCT04009668/SAP_001.pdf